CLINICAL TRIAL: NCT03030521
Title: The Roles of Intraluminal Pressure and the Dilation of Tunica Media in the Development of Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-P-011
Record Dates: First submitted 2017-01-13; First posted 2017-01-25 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- experimental group: In this group, the specimen of aortic wall is bound by a band to restrict its dilation in the fourth step of the aortic delamination test.
  Interventions: Diagnostic Test: the aortic delamination test
- control group: In this group, the specimen of aortic wall is not bound by a band to restrict its dilation in the fourth step of the aortic delamination test.
  Interventions: Diagnostic Test: the aortic delamination test

INTERVENTIONS:
Diagnostic Test: the aortic delamination test — The aortic delamination test will be performed in the dissected tissue of all patient. The processes of this test has been descripted in the summary.

SUMMARY:
Aortic dissection is defined as the separation of aortic medial lamellae. It is unknown why some aortic dissection are limited in extent while other aortic dissection extend extensively. The investigators hypothesize that the medial layers are separated as a result of the uneven dilation and dislocation of the inner and outer layers, and if this hypothesis is ture, dilation is necessary to the development of aortic dissection. In this study, an in vitro experiment was performed to test whether dilation is essential to the development of aortic dissection.

Participants will be recruited from patients with aortic repair surgery in Wuhan Asian Heart Hospital. A piece of aortic wall will be dissected to reconstruct aorta during operation. Firstly, the dissected aortic wall is sampled for routine pathological examination. Secondly, the remaining tissue is cut into a 2cm by 2cm sheet, then an incision was made on the inner surface of the tissue sheet. The outer 0.5mm media will not be incised. Thirdly, the tissue sheet is used to seal a hole in a syringe with the incision faced inside, and tissue sheet of the experimental group was bound by a band to restrict its dilation in the next step. Fourthly, the syringe is filled with blue stain, and a mechanical test is performed. Fifthly, for the experimental group, the band is removed, and the syringe is filled with red stain. The mechanical test is performed again. Finally, the tissue sheet is released and cut into several parts to show whether the inner and outer media layers are separated by the blue stain or the red stain.

DETAILED DESCRIPTION:
The mechanical test: the syringe's pressure will increase gradually to a target level, and then decrease gradually to 0 Mpa, and this process is repeated for about 60 times.

ELIGIBILITY:
Inclusion Criteria:

* patients with aortic repair surgery.

Exclusion Criteria:

* the dissected aortic wall is not big enough to be cut into a 2cm by 2cm sheet after routine pathological examination.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult patients with aortic repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
The number of patients with a positive result of the aortic delamination test | 1 month
  whether the inner and outer media layers are separated by the blue stain or the red stain.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlu Zhang, MD, Study Chair — Wuhan Asia Heart Hospital
Locations (1):
- Wuhan Asia Heart Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No
The investigators will not share participant data with other researchers.